CLINICAL TRIAL: NCT03403972
Title: A Clinical Trial to Evaluate the Effects of the Environmental Change in Intestine by Antibiotics on the Pharmacokinetic Characteristics of Simvastatin in Healthy Male Volunteers
Brief Title: Evaluate the Effects of the Environmental Change in Intestine by Antibiotics on the Pharmacokinetic Characteristics of Simvastatin in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, SeungHwan Lee, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MBSVT_PK
Record Dates: First submitted 2017-10-15; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Simvastatin Pharmacokinetics and Gut Microbiome
Keywords: pharmacokinetics; simvastatin; vancomycin; gut microbiome
MeSH Terms: interventions — Vancomycin; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Group (Experimental): Intervention: vancomycin 500 mg tid for 7 days (Vancozin 250 mg capsule)
  Interventions: Drug: Vancomycin 250Mg Capsule

INTERVENTIONS:
Drug: Vancomycin 250Mg Capsule — Investigators will compare simavastatin pharmacokinetics before and after the vancomycin PO multiple administration.
  Other Names: simvastatin

SUMMARY:
This phase 1 clinical trial is to evaluate the effects of the environmental change in intestine by antibiotics on the pharmacokinetic characteristics of simvastatin in healthy male volunteers. For change of intestine environment, especially the gut microbiota, investigators will administer PO vancomycin for 7 days, tid.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 Y to 50 Y at the screening
* Body weight over 55 kg and BMI should be between 18.0 to 25.0 kg/m2
* Informed consent will be taken before all the procedures from volunteers
* SLCO1B1 genotype is *1/*1 when screening

Exclusion Criteria:

* No significant disease history or ongoing disease
* Allergic to simvastatin and vancomycin, or similar affiliation drug for simvastatin or vancomycin
* MDRD eGFR less than 60 mL/min/1.73m2
* Total cholesterol, LDL, TG is higher than 1.5 times more than upper normal limit at the screening
* HDL less than 35 mg/dL at the screening
* Positive HBV or HIV or HCV
* Who is administering or going to administer CYP3A4 inihibitor drug
* Other clinically significant situation under doctor's opinion

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-01-11 (Actual); Study Completion 2018-01-11 (Actual)

PRIMARY OUTCOMES:
Compare the maximum plasma concentration (Cmax) | vancomycin PO will administered for 7 days
  Compare the maximum plasma concentration (Cmax) of simvastatin before and after vancomycin PO treatment.
Compare the area under the time-plasma concentration curve (AUC) | vancomycin PO will administered for 7 days
  Compare the area under the time-plasma concentration curve (AUC) of simvastatin before and after vancomycin PO treatment.

SECONDARY OUTCOMES:
Explore the gut microbiome species change | vancomycin PO will administered for 7 days
  Explore how the gut microbiome species change after vancomycin multiple dosing for 7 days

CONTACTS AND LOCATIONS:
Overall Officials: SeungHwan Lee, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital Clinical Trial Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Investigators have no plan to share individual participant data.